CLINICAL TRIAL: NCT03513224
Title: The Use of an Electronic Medication Administration-monitoring Device to Improve Medication Adherence and Reduce Medication Regimen Complexity in Community Dwelling Seniors: A Prospective Pilot Study
Brief Title: The eDosette Pilot Study
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: McMaster University (Other)
Responsible Party: Principal Investigator, Henry Siu, Assistant Professor, McMaster University
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Health Services Research
Other Study IDs: CAT2015-25
Record Dates: First submitted 2018-04-19; First posted 2018-05-01 (Actual); Last update posted 2018-05-01 (Actual); Status verified 2018-04

CONDITIONS: Medication Adherence
MeSH Terms: conditions — Medication Adherence

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- eDosette (Experimental)
  Interventions: Other: eDosette

INTERVENTIONS:
Other: eDosette — The eDosette is an internet-enabled, medication administration monitoring unit that has been previously tested for feasibility in older adults. The eDosette was designed to be compatible with different types of weekly medication blister packs and dosettes, and monitors medication-taking behaviour in a patient's home. The eDosette securely transmits this information to a secure server where the information is converted to individual medication administration records. Patients can also use the eDosette to notify their primary care team of potential medication side effects.

SUMMARY:
Medication non-adherence can lead to serious health issues for older adults. This study is a four week study in older adults using a new device, the eDosette, which dispenses and records how one takes their medications, and subsequently makes this information available to the primary care team by the internet. This study aims to show that the eDosette can report how well a group of older adults living independently in the community are taking their medications (e.g. "medication adherence"). This study hopes to show that the eDosette intervention could play a role in medication adherence by improving conversations between older adults and primary care.

ELIGIBILITY:
Inclusion Criteria:

* age 65 and over
* taking five or more medications (including supplements)
* using or willing to use a blister pack or dosette
* currently managing their medications independently
* living independently
* English speaking

Exclusion Criteria:

* a documented diagnosis of mild cognitive impairment or dementia
* living in any form of assisted living facility
* currently palliative
* currently deemed medically unstable by their primary care team

Min Age: 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Older Adult
Enrollment: 57 (Actual)
Dates: Start 2016-09-01 (Actual); Primary Completion 2017-08-31 (Actual); Study Completion 2017-12-31 (Actual)

PRIMARY OUTCOMES:
Four-week medication adherence rate | 4 weeks
  Each participant's observed medication adherence for the entire study was calculated by dividing the total medication doses taken correctly by the total doses in the study. The numerator, total medication doses taken correctly is calculated by subtracting from the total doses any missed or late doses as determined by the eDosette. Missed doses is defined as any dose still present on image data after the next daily scheduled dose time); late doses is defined as any dose taken outside the two-hour time window of the average time of dose administration - e.g. 08h00-10h00 for a 09h00 average dose time. The denominator, total doses, was defined as the total number of pills prescribed for a patient to take during the study.

SECONDARY OUTCOMES:
Thematic content of pharmacist-participant discussion during the study | 4 weeks
  Retrospective chart reviews were performed to extract content on these discussions.
Frequency of medication changes noted | 4 weeks
  Retrospective chart reviews were performed to extract content on these changes.
Change in MRCI score | 4 weeks
  Medication Regimen Complexity Index (MRCI) were calculated at baseline and 4 weeks by the pharmacist based on medication listed obtained from dispensing pharmacies.
Participant feedback | 4 weeks
  An exit-feedback survey was administered asking participants to rank their experience with the eDosette. The survey also asked participants to identify the three best and worst aspects of the eDosette.

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Siu HY, Mangin D, Howard M, Price D, Chan D. Developing and testing an electronic medication administration monitoring device for community dwelling seniors: a feasibility study. Pilot Feasibility Stud. 2017 Feb 1;3:5. doi: 10.1186/s40814-016-0118-3. eCollection 2017. PMID 28168041